CLINICAL TRIAL: NCT07172425
Title: An Open-Label, Randomised, Crossover Study to Investigate the Feasibility of Nitrate Fortification in Commonly Consumed Foods for Regulating Nitric Oxide Metabolism in Healthy Individuals
Brief Title: Evaluation of Adding Nitrate Into Foods for Regulating Nitric Oxide Bioavailability in Healthy Individuals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 180233; 10127157 (Other Grant/Funding Number: Innovate UK & BBSRC)
Record Dates: First submitted 2025-09-01; First posted 2025-09-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers; Nitric Oxide; Vascular Function
Keywords: Blood pressure; Oral microbiome profiling; Nitric oxide bioavailability; Inorganic nitrate fortification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Nitrate-fortified biscuits (NFB) (Experimental): Biscuits were fortified with 4 mmol of inorganic potassium nitrate, an amount within the acceptable daily intake (ADI) range.
  Interventions: Dietary Supplement: Inorganic potassium nitrate-fortified biscuits supplementation
- Arm 2: Nitrate-fortified cereal bar (NFCB) (Experimental): A cereal bar was fortified with 4 mmol of inorganic potassium nitrate, an amount within the acceptable daily intake (ADI) range.
  Interventions: Dietary Supplement: Inorganic potassium nitrate-fortified cereal bar supplementation
- Arm 3: Nitrate-fortified porridge (NFP) (Experimental): Porridge was fortified with 4 mmol of inorganic potassium nitrate, an amount within the acceptable daily intake (ADI) range.
  Interventions: Dietary Supplement: Inorganic potassium nitrate-fortified porridge supplementation

INTERVENTIONS:
Dietary Supplement: Inorganic potassium nitrate-fortified biscuits supplementation — Four millimoles of inorganic potassium nitrate, within the acceptable daily intake (ADI), were added to commonly consumed oat-based products (biscuits). During the trial, participants will receive nitrate-fortified biscuits as a single-day acute supplementation.
  Arms: Arm 1: Nitrate-fortified biscuits (NFB)
Dietary Supplement: Inorganic potassium nitrate-fortified cereal bar supplementation — Four millimoles of inorganic potassium nitrate, within the acceptable daily intake (ADI), were added to commonly consumed oat-based products (cereal bar). During the trial, participants will receive nitrate-fortified cereal bar as a single-day acute supplementation.
  Arms: Arm 2: Nitrate-fortified cereal bar (NFCB)
Dietary Supplement: Inorganic potassium nitrate-fortified porridge supplementation — Four millimoles of inorganic potassium nitrate, within the acceptable daily intake (ADI), were added to commonly consumed oat-based products (instant porridge). During the trial, participants will receive nitrate-fortified porridge as a single-day acute supplementation.
  Arms: Arm 3: Nitrate-fortified porridge (NFP)

SUMMARY:
Inorganic nitrate, found in leafy green vegetables and beetroot, can help lower blood pressure and support heart health. Early experimental work has suggested that dietary nitrate supplementation, in the form of beetroot juice or potassium nitrate capsules, can reduce blood pressure and improve endothelial function. Consequently, concentrated nitrate supplements like beetroot juice have become popular. However, these supplements can be expensive, high in sugar, and not to everyone's taste. Since more than three-quarters of adults with high blood pressure live in low- and middle-income countries, it is important to find safe, affordable ways to add nitrate to commonly eaten foods.

The team at Queen Mary University of London has been developing nitrate-fortified products that may be more appealing to a wider population. With support from the food manufacturer Reading Scientific Services Ltd. (RSSL), they have successfully added nitrate to three oat-based products: cereal bar, porridge, and biscuits.

This study aims to explore whether adding nitrate to commonly eaten foods can improve nitric oxide levels in the body and help lower blood pressure in healthy volunteers. Participants will receive the three nitrate-fortified food products in a randomised, crossover design. Nitrate and nitrite concentrations in biological samples, along with blood pressure, will be measured before and at multiple time points after supplementation with the nitrate-fortified products.

DETAILED DESCRIPTION:
Whether adding nitrate to commonly eaten foods can improve nitric oxide levels in the body and help lower blood pressure in healthy volunteers will be investigated.

Design: An open-label, randomised, crossover trial. Target population: Thirty healthy participants (15 males and 15 females) will be recruited.

Experimental intervention: Equal numbers of healthy male and female volunteers, aged 18-60 years, will be recruited. Following recruitment, participants will attend the clinical centre on seven occasions. At baseline, clinic blood pressure will be measured, and plasma, urine, and saliva samples will be collected. Participants will then receive one of the three nitrate-fortified food products according to the randomisation plan.

Clinic blood pressure will be measured at 1, 2, 3, and 4 hours post-supplementation. Blood samples will be collected at 0.5, 1, 1.5, 2, 2.5, 3, and 4 hours; urine at 4 hours; and saliva at 3 and 4 hours. At 24 hours post-supplementation, participants will return to the clinical centre for repeat blood pressure measurement and collection of blood, urine, and saliva samples. All human biological samples will be stored for subsequent determination of nitrate and nitrite concentrations.

If participants receive nitrate-fortified biscuits during one visit, they will be given either nitrate-fortified porridge or a cereal bar at the following visits, according to the randomisation plan. All participants will eventually receive all three nitrate-fortified food products, each providing approximately 4 mmol nitrate, an amount within the Acceptable Daily Intake (ADI) range.

The study will be conducted at the Clinical Research Centre at the William Harvey Research Institute, Queen Mary University of London.

Analysis: A two-way repeated measures ANOVA will be used to analyse the differences in [NO3-], [NO2-] in plasma, urine, and saliva, plasma [cGMP] across time and between different NO3--fortified foodstuffs (cereal bar, porridge, and biscuits) and clinic BP. Matching the objectives of comparing the changes in measures following the ingestion of the three food products, the description of the analysis will initially focus on the difference between the three food products and so post-hoc tests (accounting for multiple comparisons) will initially focus on comparing measures at each timepoint.

The acceptability of the three different NO3--fortified food products will be analysed using Friedman tests. As this is a crossover study, checks will be conducted for period effect and carry-over effect as part of the statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteer.
2. Aged ≥18 years and ≤ 60 years.
3. Willing to provide informed consent.
4. Able to understand and comply with protocol requirements, instructions, and stated restrictions.

Exclusion Criteria:

A volunteer will not be eligible for inclusion in this study if any of the following criteria are met:

1. Unwilling to provide consent.
2. People with chronic health conditions requiring medication.
3. Pregnant females, or those with a possibility of being pregnant.
4. History of hypertension and /or diabetes.
5. History of any serious illnesses, including recent infections or trauma.
6. History of symptomatic coronary artery disease, stroke, or other known atherosclerotic diseases.
7. People who will commence or who are likely to commence treatment with non-steroidal anti-inflammatory drugs (NSAIDs) other than aspirin, from screening until study completion.
8. Self-declared alcohol or drug abuse within the past 6 months.
9. Three-month prior history of regular alcohol consumption exceeding an average weekly intake of > 28 units (or an average daily intake of greater than 3 units) for males, or an average weekly intake of > 21 units (or an average daily intake of greater than 2 units) for females. One unit is equivalent to a half pint (284mL) of beer/lager; 25mL of spirits, or 125mL of wine.
10. Taking systemic medication (other than the oral contraceptive pill).
11. Recent (within 2 weeks) self-reported use of mouthwash or tongue scrapers.
12. Recent (within 2 weeks) or current antibiotic use.
13. Recent (within 1 week) use of NO3- or NO2- supplements.
14. History, or recent treatment of (within the last 3 months) for any oral condition (excluding caries), including gingivitis, periodontitis and halitosis.
15. History of, or recent treatment for, any blood-borne infectious disease such Hepatitis B or C virus, or HIV.
16. Current smokers (including vaping) or have smoked within the last 6 months.
17. Diagnosis of rheumatoid arthritis, connective tissue disorders, and other conditions known to be associated with chronic inflammation (e.g., Inflammatory Bowel Disease).
18. People who have donated more than 500mL of blood within 56 days prior to the study commencement.
19. Known allergy to celery, gluten, crustaceans, eggs, lupin, milk, mustard, peanuts, sesame, soybeans, tree nuts, oats, palm oil, sugar, cranberries, sunflower oil, invert syrup, sodium bicarbonate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
To investigate and compare the changes of NO3- and NO2- concentrations in plasma following the ingestion of three different NO3--fortified foodstuffs: cereal bar, porridge, and biscuits. | Up to 1 year
  Mean Plasma NO3- and NO2- concentrations at baseline, 0.5-, 1-, 1.5-, 2-, 2.5-, 3-, 4-, and 24-hours post-ingestion of the three NO3--fortified foodstuffs as well as area under the curve (AUC) across the 24 hours.

SECONDARY OUTCOMES:
To investigate and compare the changes of NO3- and NO2- concentrations in other human biological samples, such as saliva and urine, following the ingestion of the three different NO3--fortified foodstuffs. | Up to 1 year.
  1. Mean NO3- and NO2- concentrations in saliva at baseline, 3-, 4-, and 24-hours post-ingestion of the three NO3--fortified foodstuffs as well as AUC across the 24 hours.
  2. Mean NO3- and NO2- concentrations in urine at baseline, 4-, and 24-hours post-ingestion of the three NO3--fortified foodstuffs.
  3. The AUC of the NO3- and NO2- across the 24 hours.
To investigate and compare the changes in cGMP concentration in plasma following the ingestion of the three different NO3--fortified foodstuffs. | Up to 1 year.
  1. Mean plasma cGMP concentration at baseline and at 3 hours post-ingestion of the three NO3--fortified foodstuffs.
  2. The change at 3 hours from baseline plasma cGMP concentration.
To assess participants' acceptability of the three different NO3--fortified food products. | Final laboratory visit (assessed at this time).
  Participants' acceptability of the three different NO₃--fortified food products will be assessed through a food sensory test.
To investigate and compare the blood pressure-lowering effects of the three different NO3--fortified foodstuffs. | Up to 6 months.
  1. Mean blood pressure at baseline, 1-, 2-, 3-, 4-, and 24-hours post-ingestion of the three NO3--fortified foodstuffs.
  2. The AUC of the blood pressure across the 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Ahluwalia, BSc PhD, Study Director — Queen Mary University of London
Locations (1):
- The William Harvey Research Institute, Centre for Cardiovascular Medicines and Devices, Queen Mary University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghosh SM, Kapil V, Fuentes-Calvo I, Bubb KJ, Pearl V, Milsom AB, Khambata R, Maleki-Toyserkani S, Yousuf M, Benjamin N, Webb AJ, Caulfield MJ, Hobbs AJ, Ahluwalia A. Enhanced vasodilator activity of nitrite in hypertension: critical role for erythrocytic xanthine oxidoreductase and translational potential. Hypertension. 2013 May;61(5):1091-102. doi: 10.1161/HYPERTENSIONAHA.111.00933. Epub 2013 Apr 15. PMID 23589565
- [Background] Rathod KS, Mathur A, Shabbir A, Khambata RS, Lau C, Beirne AM, Chhetri I, Ono M, Belgaid DR, Massimo G, Ramasamy A, Tufaro V, Jain AK, Poulter N, Falaschetti E, Jones DA, Garcia-Garcia HM, Bourantas C, Learoyd A, Warren HR, Ahluwalia A. The NITRATE-OCT study-inorganic nitrate reduces in-stent restenosis in patients with stable coronary artery disease: a double-blind, randomised controlled trial. EClinicalMedicine. 2024 Oct 18;77:102885. doi: 10.1016/j.eclinm.2024.102885. eCollection 2024 Nov. PMID 39469537
- [Background] Kapil V, Khambata RS, Robertson A, Caulfield MJ, Ahluwalia A. Dietary nitrate provides sustained blood pressure lowering in hypertensive patients: a randomized, phase 2, double-blind, placebo-controlled study. Hypertension. 2015 Feb;65(2):320-7. doi: 10.1161/HYPERTENSIONAHA.114.04675. Epub 2014 Nov 24. PMID 25421976
- [Background] Kapil V, Milsom AB, Okorie M, Maleki-Toyserkani S, Akram F, Rehman F, Arghandawi S, Pearl V, Benjamin N, Loukogeorgakis S, Macallister R, Hobbs AJ, Webb AJ, Ahluwalia A. Inorganic nitrate supplementation lowers blood pressure in humans: role for nitrite-derived NO. Hypertension. 2010 Aug;56(2):274-81. doi: 10.1161/HYPERTENSIONAHA.110.153536. Epub 2010 Jun 28. PMID 20585108